CLINICAL TRIAL: NCT06143514
Title: A Post-marketing Study Evaluating the Presence and Concentration of BRIUMVI™ in Breast Milk (PROVIDE)
Brief Title: A Study Evaluating the Presence and Concentration of BRIUMVI™ (Ublituximab) in Breast Milk
Acronym: PROVIDE
Status: Recruiting | Type: Observational
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TG1101-RMS405
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Breast Milk Collection: Breast milk will be collected of participants with relapsing forms of multiple sclerosis (RMS) who are receiving BRIUMVI™ therapeutically for up to 24 hours to determine concentration of BRIUMVI™ in milk samples.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The primary objective of the lactation study is to characterize the presence and concentration of BRIUMVI™ in breast milk among breastfeeding participants who receive BRIUMVI™ therapeutically for the treatment of relapsing forms of multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

Maternal Criteria:

* Participant has independently decided to be treated with BRIUMVI™ prior to providing consent to participate in the study
* Diagnosis of RMS, to include clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), and active secondary progressive multiple sclerosis (SPMS)
* Willing to breastfeed or pump regularly during the study period to maintain milk supply and exclusively pump breast milk for the 24-hour period of breast milk collection Day 1 post IV dose
* Plans to continue feeding infant breast milk at least throughout the duration of the study and is not weaning

Infant Criteria:

* Gestational age at delivery ≥35 weeks
* Birthweight > 10th percentile
* Weight > 10th percentile as reported by the mother at the time of enrollment

Exclusion Criteria:

Maternal Criteria:

* Any active infection or other condition that would prevent the individual from breastfeeding
* History of breast implants, breast augmentation, or breast reduction surgery that significantly impacts breastfeeding or collection of milk from 1 or both breasts
* History of mastectomy
* Evidence of mastitis or any other significant active infection at Day 1 (pre-dose) that would prevent collection of milk from one or both breasts
* Current use of drugs known to transfer to the breast milk and with established or potential deleterious effects for the infant, including but not limited to aspirin (risk of Reye's syndrome), tetracyclines or fluoroquinolones

Infant Criteria:

- Any abnormality noted or clinically significant medical condition, including cardiac, pulmonary, and liver disease, glucose instability, or active infection at the time of screening that, in the opinion of the investigator, may make implementation of the protocol or interpretation of the trial difficult or would put the infant at risk by participating in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study population is restricted to breastfeeding participants.
Study Population: The study population will include breastfeeding individuals with RMS who are exposed to BRIUMVI™.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Milk Concentration-time Curve from Time 0 to Infinity (AUC0-inf) of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
Area Under the Milk Concentration-time Curve from Time 0 to the Last Measurable Observed Concentration (AUC0-last) of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
Area Under the Milk Concentration-Time Curve from Time 0 to 24 Hours Post-Dose (AUC0-24) of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
Maximum Observed Milk Concentration of BRIUMVI™ (Cmax) | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
Observed Milk Concentration of BRIUMVI™ at End of Dosing Interval (Ctrough) of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and at exit Day 90
Time of Cmax (Tmax) of BRIUMVI™ in Milk | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90

SECONDARY OUTCOMES:
Amount Excreted (Ae) of BRIUMVI™ in Milk | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
  Total amount of drug excreted in milk (mg) as: Σ(total drug concentration in each milk collection x milk volume in each milk collection)
Fraction of Dose Excreted (Fe) in Milk of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
  Fraction of dose excreted in milk calculated as Ae/Administered dose
Infant Dose (ID) of BRIUMVI™ | Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and at exit Day 90
  Infant dose = Ʃ drug concentration in each milk collection multiplied by the expressed milk volume in each milk collection.
Relative Infant Dose (RID) of BRIUMVI™ | Predose Day 1 and at multiple timepoints Post-dose Day 1, Day 2, Day 3, Day 7, Day 10, Day 14, Day 28, Day 60 and Day 90
  Relative infant dose = infant dose milligrams/kilograms (mg/kg)/ [Maternal Dose (mg)/Maternal Bodyweight (kg)] multiplied by 100
Number of Infants with Adverse Events | From the signing the inform consent form up to approximately 3 months after the index infusion

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - PROVIDE Virtual Research Coordination Center, San Francisco, California
  - PROVIDE Virtual Research Coordination Center, Smyrna, Georgia
  - PROVIDE Virtual Research Coordination Center, Wilmington, North Carolina
  - PROVIDE Virtual Research Coordination Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No